CLINICAL TRIAL: NCT03983083
Title: Health and Energy Through Active Living Every Day After Cancer: The HEALED Pilot Intervention for Cancer Survivors in CPS-3
Brief Title: Health and Energy Through Active Living Every Day (HEALED) After Cancer Pilot Intervention for Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Erika Rees-Punia, Post-Doctoral Fellow, American Cancer Society, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HEALED_CPS3
Record Dates: First submitted 2019-06-05; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Cancer; Quality of Life; Fatigue
Keywords: physical activity; sedentary behavior
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Aspects of the HEALED intervention are based on various components of successful interventions for breast cancer survivors and older adults, NCI funding priorities, CPS-3 survivor preferences discussed in prior focus groups and survivorship research from other cohorts. As such, HEALED participants will receive monthly motivational e-mails, based on prior studies of the most effective delivery time intervals for interventions involving cancer survivors, with links to a web-based platform which will provide: physical activity information (largely consisting of publicly available evidence-based resources), at-home exercise demonstrations/videos for survivors of all fitness levels, personal survivor stories, physical activity/sitting recommendations (based on National Guidelines and ACS guidelines for survivors), positive messaging, a space for SMART goal setting, a platform for physical activity tracking, a discussion board, etc.
  Interventions: Behavioral: Physical activity
- Wait-list control (No Intervention): Wait-listed control group will be instructed to continue behavior "as-usual". They will receive access to the HEALED website at the end of the 12-week intervention period.

INTERVENTIONS:
Behavioral: Physical activity — Access to website created to teach cancer survivors to live more active lives, with monthly email reminders/website updates. Intervention participants will also receive exercise bands for at-home resistance training.
  Arms: Intervention

SUMMARY:
The proposed pilot study will test the acceptability, feasibility, and safety of a twelve-week, two-arm randomized control intervention embedded within the Cancer Prevention Study-3 (CPS-3), a prospective cohort study of cancer incidence and mortality initiated by the American Cancer Society. The proposed Health and Energy through Active Living Every Day (HEALED) intervention is intended for survivors of a cancer with a 5-year survival (at Stage I and II) of at least 65% that has a strong level of evidence for association with physical inactivity according to the 2018 PA Guidelines Advisory Committee Report (breast, colon, endometrium, kidney, and bladder). In line with social cognitive theory behavior change techniques, participants will be provided information and skills necessary to be more physically active and less sedentary after a cancer diagnosis. New materials will be disseminated monthly through a website open only to participants, and include: at-home exercise demonstration videos, research news, discussion boards, success stories, infographics for exercise recommendations, etc. This intervention will add to the very minimal evidence base for PA interventions for diverse cancer survivors in a cost-effective manner.

DETAILED DESCRIPTION:
The Health and Energy through Active Living Every Day (HEALED) after cancer pilot study is a randomized consent, parallel assignment twelve-week physical activity behavioral intervention. HEALED is intended for survivors of a cancer with a 5-year survival (at Stage I and II) of at least 65% that is categorized as having a strong level of evidence for association with physical inactivity according to the 2018 Physical Activity Guidelines Advisory Committee Report, which includes: breast, colon, endometrium, kidney, and bladder.(11) HEALED has a two-arm design, including an experimental group (n=50) and a wait-listed control group (n=50) which will be instructed to continue behavior "as-usual".

Participants will be recruited through the Cancer Prevention Study-3 (CPS-3). CPS-3 is a prospective cohort study of cancer incidence and mortality initiated by the American Cancer Society (ACS). Over 254,000 CPS-3 participants aged 30 to 65 years with no history of cancer (except for basal or squamous cell skin cancer) completed a baseline survey at enrollment and are sent repeat surveys every three years to update exposure information.(17) All CPS-3 participants will be followed up for cancer incidence and mortality from any cause for at least 20 years. Between enrollment and 2015, there were over 6100 cancer cases in the CPS-3 cohort.

Eligibility for HEALED will be determined based on existing data from CPS-3 2015 and 2018 surveys. Inclusion criteria require: 1) response to 2018 CPS-3 English survey, 2) a self-reported pre- or postmenopausal breast, colon, endometrium, kidney, or bladder cancer, 3) an e-mail address on record, and 4) less than 150 minutes MVPA/week and/or no strength training reported on 2018 survey. Participants will be excluded if they: 1) are not community-dwelling, 2) are not able to walk, or 3) are currently undergoing treatment for a cancer recurrence.

Participants will be invited via email. Based on the CPS-3 physical activity sub-study, in which participants were required to wear an accelerometer for two seven-day periods and complete four seven-day diaries over a one-year period, a 20% response rate is expected. Interested participants will complete a short online screener questionnaire and provide online consent if eligible. The screening questionnaire will include items regarding stage at diagnosis and recurrence, and a physical activity readiness questionnaire (PAR-Q). Participants responding 'yes' to one or more of any of the following items will be excluded from the HEALED intervention to rule-out survivors for whom unsupervised physical activity may be unsafe: a) Has your doctor ever said that you have a heart condition and that you should only perform physical activity recommended by a doctor?, b) Do you lose your balance because of dizziness or do you ever lose consciousness?, c) Do you have a bone or joint problem that could be made worse by a change in your physical activity?, or d) Do you know of any other reason why you should not engage in physical activity? Once an eligible participant provides consent, they will be sent an accelerometer (including instructions for wear and return shipping materials) along with a 4-page survey.

ELIGIBILITY:
Inclusion Criteria:

* Response to 2018 CPS-3 English survey
* Stage I or II pre- or postmenopausal breast, colon, endometrium, kidney, or bladder cancer
* E-mail address on record
* Less than 150 minutes MVPA/week and/or no strength training reported on 2018 survey

Exclusion Criteria:

* Not community-dwelling
* Unable to walk
* Currently undergoing treatment for a cancer recurrence
* "Yes" response to PAR-Q items

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 12 weeks
  Assesses usability of the HEALED intervention website. 5-point Likert scale strongly disagree to strongly agree. The participant's scores for each question are converted to numbers 0-4, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average.
  Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking.
Physical activity | 12 weeks
  Objectively-measured moderate-vigorous physical activity, light physical activity, and sedentary time
Number of exercise-related adverse events (self-reported musculoskeletal injuries, falls, etc.) | 12 weeks
  Safety of HEALED intervention

SECONDARY OUTCOMES:
Fatigue Symptom Inventory | 12 weeks
  Physical and mental fatigue, 14 items. Items use an 11-point, Likert-type scale that ranges from one fatigue-related extreme to another (lower points on the scale denote less acute problems with fatigue). A global score can be obtained for items 1-13. Question 14 is meant to provide qualitative data only.
PROMIS Sleep Disturbance (short form 6a) | 12 weeks
  Sleep disturbances and overall sleep quality, 6 items. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 6 to 30 with higher scores indicating greater severity of sleep disturbance.
University of Minnesota Cognitive Function Survey | 12 weeks
  Survey-assessed cognitive function from the Long-Term Follow-Up Study. 25 items with three-point Likert-type scale ranging from "Never a problem" to "Often a problem". Scores range from 25-75, with scores above 50 indicating issues with cognitive function (largely problem-solving).

CONTACTS AND LOCATIONS:
Locations (1):
- American Cancer Society, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rees-Punia E, Leach CR, Westmaas JL, Dempsey LF, Roberts AM, Nocera JR, Patel AV. Pilot Randomized Controlled Trial of Feasibility, Acceptability, and Preliminary Efficacy of a Web-Based Physical Activity and Sedentary Time Intervention for Survivors of Physical Inactivity-Related Cancers. Int J Behav Med. 2022 Apr;29(2):220-229. doi: 10.1007/s12529-021-09999-5. Epub 2021 May 6. PMID 33954891